CLINICAL TRIAL: NCT05552651
Title: A Single-arm, Exploratory Clinical Study of Envafolimab Combined With Chemotherapy in Neoadjuvant Therapy for Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Envafolimab Combined With Chemotherapy in Neoadjuvant Therapy for Resectable Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tao Jiang (Other)
Responsible Party: Sponsor-Investigator, Tao Jiang, Department director, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202208-20
Record Dates: First submitted 2022-09-14; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: neoadjuvant therapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — envafolimab; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab plus chemotherapy (Experimental)
  Interventions: Drug: Envafolimab; Drug: Albumin-Bound Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Envafolimab — 300mg,sc,d1,Q3W;
Drug: Albumin-Bound Paclitaxel — 130mg/m2,iv,D1,D8,Q3W
Drug: Carboplatin — AUC=5, iv,D1,Q3W

SUMMARY:
The objective is to investigate the efficacy and safety of envafolimab combined with chemotherapy for preoperative neoadjuvant therapy in patients with resectable esophageal squamous cell carcinoma

DETAILED DESCRIPTION:
This study is a single-arm, exploratory phase II clinical study. In the study, all patients with esophageal squamous cell carcinoma who meet the inclusion criteria will receive 3 cycles (21 days of 1 cycle) of neoadjuvant envolizumab combined with chemotherapy Treatment, radical surgery 4-6 weeks after completion of the last neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study, signed the informed consent form, and had good compliance;
* 18-75 years；
* ECOG 0-1；
* life expectancy of at least 3 months；
* For patients diagnosed with thoracic esophageal squamous cell carcinoma by histopathological examination of the primary tumor, the stage of esophageal cancer was clearly diagnosed as cT1b-cT2 N+ or cT3-cT4a anyN stage by CT or MRI or color Doppler ultrasound or PET-CT or ultrasonography before surgery , and evaluated by the investigator as suitable for patients treated with this study protocol.
* Not received any anti-tumor therapy in the past, including but not limited to surgery, radiotherapy, chemotherapy, immunotherapy, targeted therapy, etc. However, exploratory thoracotomy, mediastinoscopy, excisional biopsy or similar surgical procedures for definite diagnosis, staging and surgical treatment of esophageal cancer can be accepted.
* Satisfactory main organ function，laboratory test must meet the following criteria: hemoglobin (HGB) ≥90g/L, neutrophil count（ANC） ≥1.5×109/L, platelet count（PLT） ≥80×109/L, Serum creatinine（CR）≤1.5 upper normal limitation (UNL)，total bilirubin (TBil) ≤1.5 upper normal limitation (UNL), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 UNL (For patients with liver metastasis, the AST/ALT must be ≤5.0 UNL), Activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5×ULN; left ventricular ejection fraction (LVEF) ≥ 50%; thyroid stimulating hormone (TSH) within the normal range Within: if the baseline TSH exceeds the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
* The doctor's clinical judgment has sufficient organ function;
* Subjects of childbearing potential must use an appropriate method of contraception during the study period and within 120 days after the end of the study, have a negative serum pregnancy test within 7 days prior to study enrollment, and must be non-lactating subjects ；

Exclusion Criteria:

* Suffered from other malignant tumors within 5 years before the start of treatment in this study;
* Patients with tumor invading the cervical esophagus or high upper thoracic segment requiring a laryngectomy;
* Patients with a high risk of bleeding or perforation due to the obvious invasion of the tumor into the adjacent organs (aorta or trachea) of the esophageal lesion, or patients who have already formed a fistula;
* Subjects with any severe and/or uncontrolled disease;
* Poor blood pressure control (systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥ 90mmHg);
* Subjects with any severe and/or uncontrolled disease ；
* Have clinical symptoms or diseases of the heart that are not well controlled；
* Patients with past and current objective evidence of history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severely impaired lung function；
* Acute or chronic active hepatitis B (hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive patients need to be tested for hepatitis B virus (HBV) DNA, such as HBV DNA copy number ≤2×103 copies/ml or ≤200 IU/ml or below the lower limit of detection, can be enrolled. HBsAg (+) subjects should receive anti-HBV therapy throughout the study drug treatment period to avoid viral activation. For anti-HBV Subjects with HBc(+), HBsAg(-), anti-HBs(-) and HBV viral load(-) do not need to receive preventive anti-HBV treatment, but need to be closely monitored for virus reactivation;
* A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
* Poor control of diabetes (fasting blood glucose [FBG]> 10mmol/L);
* Clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction;
* Those who have received major surgical treatment, incision biopsy or obvious traumatic injury within 28 days before the start of study treatment; or have long-term unhealed wounds or fractures;
* Serious arterial/venous thrombotic events, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism, occurred within 6 months before the start of study treatment;
* Those who have a history of psychotropic substance abuse and cannot quit or have mental disorders;
* Patients who have received tumor treatment in the past;
* Subjects with uncontrolled pleural effusion, pericardial effusion or ascites (judgment by the investigator) who still need repeated drainage;
* Subjects with known central nervous system metastases and/or cancerous meningitis;
* History of vaccination with live attenuated vaccine within 14 days before the start of study treatment or planned vaccination with live attenuated vaccine during the study period;
* Active autoimmune disease requiring systemic treatment (such as the use of disease-modifying drugs, corticosteroids or immunosuppressants) within 2 years before the start of study treatment, alternative therapy (such as thyroxine, insulin, or adrenal or pituitary use) Physiological corticosteroids with insufficiency, etc.) are excluded;
* Diagnosed with immunodeficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy. (dose>10mg/day prednisone or other equivalent therapeutic hormones), and continued use within 2 weeks of the first administration;
* Those with a history of active tuberculosis;
* Within 4 weeks before the start of the study, are participating in or have participated in other clinical investigators;
* Those who have been treated with other PD-1/PD-L1 inhibitors in the past cannot be enrolled; the subjects are known to be allergic to macromolecular protein preparations, or known to be allergic to the applied drug components;
* Those who are known to be allergic to the active ingredients or excipients of the study drugs such as envolimab, nab-paclitaxel, and nedaplatin;
* According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or subjects who are considered unsuitable for enrollment for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-20 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Rate of pCR | From Baseline to primary completion date, about 6 months
  Rate of pathological complete remission

SECONDARY OUTCOMES:
Rate of MPR | From Baseline to primary completion date, about 6 months
  Rate of major pathological remission

OTHER OUTCOMES:
Rate of SAE | From Baseline to primary completion date, about 18 months
  Rate of severity Adverse Event

IPD SHARING:
Plan to Share IPD: No